CLINICAL TRIAL: NCT02566447
Title: "Solana™ Trichomonas Assay Field Study"
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TV-01-2015
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2017-08

CONDITIONS: Trichomonas Vaginalis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Trichomonas vaginalis in vaginal swabs and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Symptomatic: Subjects will be categorized by the clinician as symptomatic for Trichomonas vaginalis infection.
  Interventions: Device: Solana Trichomonas Assay Testing

INTERVENTIONS:
Device: Solana Trichomonas Assay Testing — Specimen collection of urine and/or vaginal swabs for testing

SUMMARY:
The Solana® Trichomonas Assay is an in vitro qualitative nucleic acid amplification test for the detection of Trichomonas vaginalis to aid in the diagnosis of trichomoniasis using the Helicase-Dependent Amplification (HDA) technology and the Solana instrument.

DETAILED DESCRIPTION:
This study is to establish the clinical performance of the Solana® Trichomonas Assay for the detection of Trichomonas vaginalis in vaginal swabs and urine samples as compared to a combined reference method of direct wet mount microscopy and a FDA-cleared device.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects will be recruited from the general population as they present to the clinical facility. Subjects will be categorized by the clinician as either asymptomatic or symptomatic for Trichomonas vaginalis infection.

Symptoms in women can include:

* Greenish-yellow, frothy vaginal discharge with a strong odor
* Painful urination
* Vaginal itching and irritation
* Discomfort during intercourse
* Lower abdominal pain (rare)

Exclusion Criteria:

1. The study is limited to females. Male subjects are not accepted.
2. At clinical sites informed consent, unable to understand and consent to participation; for minors this includes parent or legal guardian.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects symptomatic for Trichomonas vaginalis infection.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Trichomonas Test Result | 2 days
  Testing results will be received by testing site for current FDA cleared tests

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of North Carolina, Div. of Infectious Diseases, Chapel Hill, North Carolina
  - University of Washington in Seattle, Seattle, Washington